CLINICAL TRIAL: NCT07328477
Title: Effect of Box Breathing Technique on Anxiety, Pain, and Nausea in Patients Undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP): A Randomized Controlled Trial
Brief Title: Box Breathing for Anxiety, Pain and Nausea in ERCP Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-09-349
Record Dates: First submitted 2025-12-30; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography; Anxiety; Pain; Nausea
Keywords: Box breathing; Breathing exercises; Non-pharmacological intervention; Nursing intervention; ERCP; Anxiety management; Pain management; Nausea management
MeSH Terms: conditions — Anxiety Disorders; Pain; Nausea; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two parallel groups: an intervention group receiving box breathing in addition to standard care, and a control group receiving standard care alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Box Breathing Group (Experimental): Participants receive standard care plus box breathing training before ERCP.
  Interventions: Behavioral: Box Breathing Technique
- Control Group (No Intervention): Participants receive standard pre-procedural care only.

INTERVENTIONS:
Behavioral: Box Breathing Technique — Box breathing is a structured breathing technique consisting of four equal phases: inhalation for four seconds, breath holding for four seconds, exhalation for four seconds, and breath holding again for four seconds. The technique is taught by a nurse one day before ERCP and practiced approximately 30 minutes before the procedure.
  Arms: Box Breathing Group

SUMMARY:
This study aims to evaluate the effects of a non-pharmacological breathing technique, known as box breathing, on anxiety, pain, and nausea in adult patients undergoing endoscopic retrograde cholangiopancreatography (ERCP). ERCP is an invasive endoscopic procedure that may cause significant physical and psychological discomfort, including increased anxiety, pain, and nausea.

Participants are randomly assigned to either an intervention group receiving standard care plus box breathing training or a control group receiving standard care alone. The box breathing technique consists of four equal phases of breathing (inhale, hold, exhale, hold), each lasting four seconds. Anxiety, pain, and nausea levels are assessed before ERCP and within the first 24 hours after the procedure. The results of this study may contribute to improving patient comfort and supporting the use of simple, nurse-led interventions in clinical practice.

DETAILED DESCRIPTION:
This single-center randomized controlled trial investigates the effectiveness of the box breathing technique on anxiety, pain, and nausea in patients undergoing endoscopic retrograde cholangiopancreatography (ERCP). The study is conducted in the gastroenterology clinic of a tertiary care hospital in Turkey.

Adult patients scheduled for ERCP who meet the inclusion criteria are enrolled and randomly assigned to either the intervention group or the control group using simple randomization. Patients in the intervention group receive standard pre-procedural care in addition to structured box breathing training provided by a nurse one day before the ERCP procedure. The box breathing technique involves four equal breathing phases: inhalation for four seconds, breath-holding for four seconds, exhalation for four seconds, and breath-holding again for four seconds. Participants are reminded to practice the technique approximately 30 minutes before the procedure and are encouraged to continue its use after ERCP.

Patients in the control group receive standard care only, without breathing training. Data are collected using validated instruments. Anxiety levels are measured using the State Anxiety Inventory (STAI), pain intensity is assessed using the Visual Analog Scale (VAS), and nausea, vomiting, and retching are evaluated using the Rhodes Index. Baseline measurements are obtained before the procedure, and follow-up assessments are completed within 24 hours after ERCP.

The primary outcome of the study is the change in anxiety levels. Secondary outcomes include pain intensity and nausea severity. This study aims to provide evidence on the effectiveness of a simple, non-invasive, and nurse-led breathing intervention to improve symptom management and patient comfort during invasive endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Scheduled to undergo endoscopic retrograde cholangiopancreatography (ERCP)
* Able to communicate verbally
* Able to understand and perform the box breathing technique
* Willing to participate and provide written informed consent

Exclusion Criteria:

* Cognitive impairment or psychiatric disorders affecting cooperation
* Hearing or communication problems that prevent understanding instructions
* Use of sedative or anxiolytic medication before ERCP other than standard sedation
* Previous participation in breathing or relaxation training programs
* Emergency ERCP procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Anxiety level | From baseline (before ERCP) to within 24 hours after ERCP
  Anxiety level will be assessed using the State Anxiety Inventory (STAI). The scale consists of 20 items, with higher scores indicating higher levels of anxiety.

SECONDARY OUTCOMES:
Pain intensity | Within 24 hours after ERCP
  Pain intensity will be measured using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst possible pain).
Nausea severity | Within 24 hours after ERCP
  Nausea, vomiting, and retching will be evaluated using the Rhodes Index of Nausea, Vomiting, and Retching (INVR). Higher scores indicate greater symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is a single-center academic study and the informed consent obtained from participants did not include provisions for data sharing beyond the research team. Data are stored securely and will be used only for the purposes defined in the study protocol.